CLINICAL TRIAL: NCT06103552
Title: Building Lifestyle Options for Orthopedic Mobility: Preoperative Weight Loss and Impact on Health in People Living With Obesity Awaiting Orthopedic Procedure
Brief Title: BLOOM Forward: Investigating Weight Loss Impact on TJAC Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: LEAF Weight Loss Clinic (Unknown); The Ottawa Hospital (Other)
Responsible Party: Principal Investigator, Judy Shiau, Investigator, Ottawa Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230569-01H
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Obesity; Knee Osteoarthritis; Hip Osteoarthritis; Arthroplasty Complications
Keywords: Obesity; Body Mass Index; Weight Loss; Noncommunicable Diseases; Surveys and Questionnaires; Metabolic Disease; Arthroplasty; Osteoarthritis; Joint Diseases
MeSH Terms: conditions — Obesity; Osteoarthritis, Knee; Osteoarthritis, Hip; Weight Loss; Noncommunicable Diseases; Metabolic Diseases; Osteoarthritis; Joint Diseases

STUDY DESIGN:
Intervention Model Description: This is an open label, single arm, cohort study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Weight Loss Program Intervention (Experimental): All study participants will be assigned to the intervention arm of this trial where they will undergo the BLOOM lifestyle program for weight loss. This program is 24 weeks in duration and includes group nutrition coaching with a dietitian, regular physician appointments and access to online support materials. Participants may also choose to pursue weight loss medication or meal replacement therapy, although this is not specifically part of the BLOOM program being studied.
  Interventions: Behavioral: Building Lifestyle Options for Orthopedic Mobility (BLOOM)

INTERVENTIONS:
Behavioral: Building Lifestyle Options for Orthopedic Mobility (BLOOM) — This intervention is a lifestyle program with includes dietary coaching from a dietitian and regular doctor appointments with a bariatric medicine specialist over the course of 24 weeks.

SUMMARY:
The goal of this clinical trial is to prospectively assess the efficacy of the BLOOM program, a comprehensive weight loss dietary and lifestyle program, in a population of patients living with obesity and awaiting hip or knee surgery. The main questions it seeks to answer are:

1. Can the BLOOM program support these patients to lose up to 10% of their initial body weight?
2. Will patients continue to lose weight for the next six months after completing the program?
3. Does the BLOOM program help patients to improve their overall quality of life?

Study participants will undergo the BLOOM program, a virtual pre-operative weight management program that spans 24 weeks and is carefully supervised by medical professionals. They will be recruited at the LEAF Clinic after being referred by their primary care physician.

During the BLOOM program, they will meet with a physician (initially, then once monthly) and a dietitian (initially, and then biweekly as part of virtual group coaching). They will have access to LEAF's online learning portal. These are normal elements of the BLOOM program.

Furthermore, as part of their participation in the research study, participants will be asked to complete the following questionnaires: the Mediterranean dietary score, the Oxford Hip and Knee Questionnaire and the EQ-D5-5L quality of life assessment. They will complete these initially, and then at completion of the program and 3 and 6 months post-program. We will also collect their height and weight at these intervals.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the study, subjects must meet all the following criteria:

  1. Age ≥ 18 years old
  2. Body mass index (BMI) ≥ 35 kg/m2
  3. Have being identified as a potential orthopedic surgery candidate by the Total Joint Assessment Clinic (TJAC)
  4. Have a referral by their primary care practitioner
  5. Ready to participate actively in the program (i.e., readiness to change scale score ≥7)
  6. Acquisition of the required technology tools and skills to use the virtual platform (the BLOOM program will be conducted via virtual video conference)
  7. English comprehension at a level that allows for active participation in the program

Exclusion Criteria:

* Subjects who meet any of the following criteria are not eligible for the study:

  1. Active eating disorder
  2. Active substance use disorder
  3. Active smoking
  4. Currently or past enrollment in another weight loss program in the previous year prior to enrollment in the study
  5. Ongoing pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Weight loss | Weight will be compared from beginning of program to end of program, six months after program completion, and also monthly for months 1-5.
  The difference (in lbs and %) in weight between the admission visit and the end of the BLOOM program

SECONDARY OUTCOMES:
Weight - BMI 35-40 | Six months
  The difference (in lbs and %) in weight between the admission visit and the end of the BLOOM program for individuals with a BMI of 35-39.9
Weight - BMI 40+ | Six months
  The difference (in lbs and %) in weight between the admission visit and the end of the BLOOM program for individuals with a BMI over 40
Mediterranean Diet Score | At program start, at program completion (approx 6 months, 3 and 6 months post-program completion (total time: twelve months)
  The change in the Mediterranean Dietary Score between the initial visit and the end of the BLOOM program and 3 and 6 months after
Oxford Knee and Hip | At program start, at program completion (approx 6 months, 3 and 6 months post-program completion (total time: twelve months)
  The change in the Oxford Hip and Knee Questionnaires between the initial visit and the end of the BLOOM program and three and six months after.
EQ-5D-5L | At program start, at program completion (approx 6 months, 3 and 6 months post-program completion (total time: twelve months)
  The change in the EQ-5D-5L quality of life (QoL) score between the initial visit and the end of the BLOOM program and three and six months after.
Decision change | Twelve months
  The proportion of patients that have a change of decision for joint arthropathy.
Weight change | Twelve months
  The proportion of patients who continued to lose weight or maintained their weight 3 and 6 months after the end of the program

CONTACTS AND LOCATIONS:
Overall Officials: Judy Shiau, MD, Principal Investigator — The Ottawa Hospital

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share IPD with other researchers, nor are we seeking institutional ethical approval for such sharing.